CLINICAL TRIAL: NCT01314586
Title: Iowa State Study on Flax Lignans and Heart Health
Brief Title: Flax Lignans and Heart Health
Acronym: ISULignan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Collaborators: Archer Daniels Midland Co. (Industry)
Responsible Party: Suzanne Hendrich, PhD, University Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ADM Beneflax ISU-1
Record Dates: First submitted 2011-03-09; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; postmenopause; secoisolariciresinol diglucoside; flaxseed; lignans; enterolactone; enterodiol; serum cholesterol; LDL cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): placebo pill, diet counseling to comply with NCEP Step I diet
  Interventions: Dietary Supplement: secoisolariciresinol diglucoside-containing extract of flaxseed
- 150 mg/day Beneflax (Experimental): 2 pills taken at breakfast and dinner containing a total of 150 mg secoisolariciresinol (SDG) per day for 12 weeks
  Interventions: Dietary Supplement: secoisolariciresinol diglucoside-containing extract of flaxseed
- 300 mg/day Beneflax (Experimental): 2 pills taken at breakfast and dinner containing a total of 300 mg secoisolariciresinol (SDG) per day for 12 weeks
  Interventions: Dietary Supplement: secoisolariciresinol diglucoside-containing extract of flaxseed

INTERVENTIONS:
Dietary Supplement: secoisolariciresinol diglucoside-containing extract of flaxseed — 0, 150 or 300 mg/day as 2 pills taken at breakfast and dinner, dietary counseling to comply with NCEP Step I diet
  Other Names: Beneflax

SUMMARY:
Purpose: To demonstrate the efficacy of Beneflax™ flaxseed lignan (SDG) concentrate to lower serum cholesterol levels.

Background: Flaxseed has been studied for various health benefits in humans, including prostate health, glucose control, and cardiovascular health. Cholesterol levels and high blood pressure are known to be risk factors for cardiovascular disease. Whole flaxseed has had variable effects on serum lipid levels, perhaps a consequence of variations in the amounts of secoisolariciresinol diglucoside (SDG) found in different flax cultivars, making the study of this bioactive compound difficult.

Hypothesis: Flaxseed lignan (SDG) extract (Beneflax) significantly lowers total and LDL cholesterol. Flaxseed lignans also lower blood pressure and fasting glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Men, 40-65 yrs/old, postmenopausal women 50-65 yrs/old not > 5 yrs post menopause. All subjects were hypercholesterolemic with either total cholesterol >240 mg/dl and < 320 mg/dL or LDL cholesterol >140 mg/dl and <190 mg/dl at the screening visit.

Exclusion Criteria:

* Excluded subjects included diabetics, people being actively treated with niacins, fibrates, statins, insulin, ACE inhibitors or other cholesterol/ blood pressure pharmaceutical treatments, people who consumed large amounts of soy, flax, rye breads, pumpkin seeds, hydrolyzed milk products, sterols, and/or berries (strawberries/blueberries) or supplements aimed at cholesterol reduction such as spruce lignans, sytrinol (poly methoxylated flavanols), polycosinols, people consuming flaxseed on a regular basis.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in serum total cholesterol from baseline to 12 weeks after intervention treatments | 12 weeks
Change in serum glucose from baseline to 12 weeks after intervention treatments | 12 weeks
Change in blood pressure from baseline to end of treatment | 12 weeks

SECONDARY OUTCOMES:
Changes in serum clinical chemistry from baseline to end of treatment | 12 weeks
  serum uric acid, BUN, Na, K, Cl, Ca, P, LDH, AST, ALT, bilirubin, carbon dioxide

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Hendrich, PhD, Principal Investigator — Iowa State University
Locations (1):
- Nutrition & Wellness Research Center, Ames, Iowa, United States